CLINICAL TRIAL: NCT00124527
Title: Phase 2 Clinical Trial of Bi-weekly Dosing of Irofulven Plus Capecitabine in Patients With Anaplastic or Locally Advanced/Metastatic Differentiated Thyroid Cancer
Brief Title: Study of Irofulven Plus Capecitabine in Patients With Advanced Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IROF-019
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2008-11

CONDITIONS: Thyroid Cancer
Keywords: Irofulven, Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — irofulven; Capecitabine

INTERVENTIONS:
Drug: Irofulven + capecitabine

SUMMARY:
Irofulven is an investigational chemotherapeutic agent being studied in a variety of solid tumors. The purpose of this study is to assess the efficacy and safety of irofulven/capecitabine combination therapy in patients with anaplastic, medullary, or locally advanced/metastatic differentiated thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Cancer of the thyroid confirmed by a biopsy sample. Specific types of thyroid cancer included in this study are anaplastic, differentiated (papillary, follicular, or Hürthle cell), and medullary thyroid cancers.
* For patients with differentiated (papillary, follicular, or Hürthle cell) thyroid cancer, no more than 1 prior chemotherapy treatment is allowed.
* Measurable disease is required (at least one lesion at least 2 cm in length by conventional computed tomography (CT) techniques or at least 1 cm by spiral CT scan).
* Any prior chemotherapy or radiation therapy must be stopped at least 4 weeks before the first dose of study treatment. Prior radioiodine (I131) therapy must be stopped at least 3 (or 6) months before first dose of study treatment (depending on responsiveness to this therapy).
* Recovery from any toxic effects of prior chemotherapy, radiation therapy and surgery.
* Patients with reproductive potential must use a medically acceptable contraceptive method. Women of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* History of retinopathy.
* Serious ongoing medical or psychiatric disorder (as determined by the clinical investigator).
* External beam radiation therapy to >30% of the bone marrow at any time prior to study entry.
* Prior treatment with irofulven or capecitabine, or protracted infusion of 5-fluorouracil (5-FU) (infusion duration greater than or equal to 5 days) or other fluoropyrimidines.
* Therapeutic doses of coumarin derivatives (warfarin) 14 days prior to receiving the first dose of study treatment or during the study period.

Please note: There are additional criteria that must be met in order to be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2005-03-31 (Actual); Primary Completion 2006-08-31 (Actual); Study Completion 2006-08-31 (Actual)

PRIMARY OUTCOMES:
To determine the objective tumor response rate in patients with anaplastic, medullary, or locally advanced/metastatic differentiated thyroid cancer treated with irofulven/capecitabine combination therapy

SECONDARY OUTCOMES:
To evaluate the safety of irofulven/capecitabine combination therapy in patients with anaplastic, medullary, or locally advanced/metastatic differentiated thyroid cancer
To determine time-to-event variables of overall survival, time to disease progression, time to response, and duration of response

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - Aurora, Colorado
  - Columbus, Ohio
- Salta, Argentina
- France (3):
  - Lyon
  - Toulouse
  - Villejuif
- Lima, Peru
- Russia (2):
  - Moscow
  - Obninsk
- Kiev, Ukraine